CLINICAL TRIAL: NCT00617448
Title: Ligasure™ Versus Diathermy Haemorrhoidectomy Under Spinal or Local Anaesthesia With Ropivacaine. A Randomized Study With One Year Follow-up
Brief Title: Ligasure Versus Diathermy Haemorrhoidectomy Under Local Anesthesia
Acronym: LDHLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Viladecans (Other)
Collaborators: Fundacio per la recerca e investigació del Hospital de Viladecans (Unknown)
Responsible Party: Felip Pi Siques, Departement of Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05/0008
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Hemorrhoids
Keywords: diathermy hemorrhoids; Ligasure; randomized controlled trial; Postoperative pain; Surgical Procedure, Ambulatory; Local Anesthesia; Safety procedure long term; Day Surgery
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative | interventions — Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- I (Active Comparator): conventional diathermy haemorrhoidectomy under spinal anaesthesia
  Interventions: Procedure: diathermy haemorrhoidectomy under espinal anesthesia
- II (Active Comparator): conventional diathermy haemorrhoidectomy with local anaesthesia combined with intravenous sedation (group II)
  Interventions: Procedure: diathermy haemorrhoidectomy under local anesthesia
- III (Active Comparator): Ligasure haemorrhoidectomy under spinal anesthesia
  Interventions: Procedure: Ligasure haemorrhoidetomy under spinal anestesia
- IV (Active Comparator): Ligasure haemorrhoidectomy under local anesthesia
  Interventions: Procedure: Ligasure haemorrhoidectomy under local anesthesia

INTERVENTIONS:
Procedure: diathermy haemorrhoidectomy under espinal anesthesia — For surgery: conventional haemorrhoidectomy with diathermy (Milligan-Morgan).For anesthesia: lidocaine 2% at doses of 50-70 mg was used for spinal anaesthesia.
  Other Names: diathermy excision haemorrhoids regional; open haemorrhoidectomy; regional anesthesia
  Arms: I
Procedure: diathermy haemorrhoidectomy under local anesthesia — For surgery: conventional haemorrhoidectomy with diathermy (Milligan-Morgan). For anesthesia: pudendal nerve block, infiltration of the right and left pararectal spaces, anterior and presacral regions with ropivacaine (150 mg of ropivacaine [20 mL, 7.5 mg/mL] diluted in 50 mL of 0.9% physiological saline). Ten minutes before local anaesthesia, patients were sedated with i.v. remifentanil 0.05-0.15 μg·kg-1
  Other Names: diathermy excision haemorrhoids regional; open haemorrhoidectomy; perianal anesthetics infiltration; pudendal block
  Arms: II
Procedure: Ligasure haemorrhoidetomy under spinal anestesia — For surgery: ligasure haemorrhoidectomy For anesthesia: lidocaine 2% at doses of 50-70 mg was used for spinal anaesthesia.
  Other Names: regional anesthesia; Ligasure for prolapsed piles
  Arms: III
Procedure: Ligasure haemorrhoidectomy under local anesthesia — For surgery: haemorrhoidectomy with Ligasure For anesthesia: pudendal nerve block, infiltration of the right and left pararectal spaces, anterior and presacral regions with ropivacaine (150 mg of ropivacaine [20 mL, 7.5 mg/mL] diluted in 50 mL of 0.9% physiological saline). Ten minutes before local anaesthesia, patients were sedated with i.v. remifentanil 0.05-0.15 μg·kg-1
  Other Names: Ligasure for prolapsed piles; Pudendal block
  Arms: IV

SUMMARY:
The objective of this prospective randomised trial was to compare the short- and long-term efficacy of conventional diathermy haemorrhoidectomy versus Ligasure™ diathermy, and to assess the short-term outcome of each procedure performed either under spinal anaesthesia or local anaesthesia with pudendal block with ropivacaine combined with intravenous sedation.

We think, Ligasure haemorrhoidectomy under local anesthesia can be performed as day-case procedure and with equal results at long-term than conventional diathermy (considered goal standar of haemorrhoidectomy).

DETAILED DESCRIPTION:
Seventy-four consecutive patients with a long-standing history of symptomatic grade III or IV haemorrhoids were assigned randomly by means of a computer-generated list to conventional diathermy haemorrhoidectomy under spinal anaesthesia (group I); conventional diathermy haemorrhoidectomy with local anaesthesia combined with intravenous sedation (group II); Ligasure™ under spinal anaesthesia (group III) and Ligasure™ with local anaesthesia combined with intravenous sedation (group IV). Allocations were sealed in opaque numbered envelopes. All patients were operated on electively and by the same surgical team (two colorectal surgeons) and variables were collected after operation by an independent observer who was unaware of the operation performed.

The intraoperative time was measured. Intraoperative and early (within the first 48 h) postoperative complications associated with the surgical procedure and complications related to the anaesthetic technique (headache, vomiting, nausea, acute urinary retention, bleeding and hypotension) were recorded. A 100-mm visual analogue scale (VAS) was used to assess the intensity of pain, which was measured at 2, 6 and 24 hours postoperatively and during the first bowel movement. Seven days after surgery, patients were contacted by phone and the following data were recorded: VAS score at rest and during bowel movements, bleeding (categorised as 0 = none, 1 = occasional with defecation, 2 = with each defecation, 3 = with and without defecation) and pruritus (categorised as 0 = none, 1 = occasional, 2 = frequent) and tenesmus (categorised as 0 = none, 1 = occasional, 2 = frequent). These variables were collected at 4 and 12 months after operation by an independent observer who was unaware of the operation performed. Clinical evaluation at 1 year included relapse, continence according to the incontinence score system of Jorge and Wexner19, anal stenosis, presence of skin tags, patient's degree of satisfaction (where 0 corresponded to a unsatisfactory result and 10 an excellent result) and days of sick leave.

ELIGIBILITY:
Inclusion Criteria:

* patients with a long-standing history of symptomatic grade III or IV haemorrhoids

Exclusion Criteria:

* previous anal surgery, concomitant anal disease (fissure, fistula, incontinence and inflammatory bowel disease), use of anticoagulants or analgesics, known hypersensitivity to local anaesthetics and the inability to give written informed consent.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2005-05; Primary Completion 2006-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
all cause morbility within the first 7 days after surgery (consequence of surgery and anesthesia) and results sintomatology since 12 months | at 2, 6, 24 horus, 7 days, 4 and 12 monts after surgery

SECONDARY OUTCOMES:
intraoperative time, postoperative complications, pain (VAS), bleeding, pruritus and tenemus, continence ( score system of Jorge and Wexner), anal stenosis, presence of skin tags, degree of satisfaction and days of sick leave. | Intraoperative, at 2,6,24 hours and 7 days after surgery and 4 and 12 monts after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pi F Siques, Professor, Principal Investigator — Barcelona university of Medicine (Departement Ciencies Cliniques)
Locations (1):
- Hospital de Viladecans (Departement of surgery: coloproctology), Viladecans, Barcelona, Spain

REFERENCES:
- [Result] Jayne DG, Botterill I, Ambrose NS, Brennan TG, Guillou PJ, O'Riordain DS. Randomized clinical trial of Ligasure versus conventional diathermy for day-case haemorrhoidectomy. Br J Surg. 2002 Apr;89(4):428-32. doi: 10.1046/j.0007-1323.2002.02056.x. PMID 11952582
- [Result] Palazzo FF, Francis DL, Clifton MA. Randomized clinical trial of Ligasure versus open haemorrhoidectomy. Br J Surg. 2002 Feb;89(2):154-7. doi: 10.1046/j.0007-1323.2001.01993.x. PMID 11856126
- [Result] Peters CJ, Botterill I, Ambrose NS, Hick D, Casey J, Jayne DG. Ligasure trademark vs conventional diathermy haemorrhoidectomy: long-term follow-up of a randomised clinical trial. Colorectal Dis. 2005 Jul;7(4):350-3. doi: 10.1111/j.1463-1318.2005.00817.x. PMID 15932557
- [Result] Basdanis G, Papadopoulos VN, Michalopoulos A, Apostolidis S, Harlaftis N. Randomized clinical trial of stapled hemorrhoidectomy vs open with Ligasure for prolapsed piles. Surg Endosc. 2005 Feb;19(2):235-9. doi: 10.1007/s00464-004-9098-0. Epub 2004 Dec 2. PMID 15573239
- [Result] Masoni L, La Torre F, Otti M, Pascarella G, Gasparrini M, Riso V, Cottini F, Montori A. [Hemorrhoidectomy with ropivacaine (Naropin) local anesthesia. Preliminary experience]. Minerva Chir. 2000 May;55(5):383-7. Italian. PMID 10953578
- [Result] Lohsiriwat D, Lohsiriwat V. Outpatient hemorrhoidectomy under perianal anesthetics infiltration. J Med Assoc Thai. 2005 Dec;88(12):1821-4. PMID 16518980
- [Result] Vinson-Bonnet B, Coltat JC, Fingerhut A, Bonnet F. Local infiltration with ropivacaine improves immediate postoperative pain control after hemorrhoidal surgery. Dis Colon Rectum. 2002 Jan;45(1):104-8. doi: 10.1007/s10350-004-6121-4. PMID 11786772
- [Result] Kim J, Lee DS, Jang SM, Shim MC, Jee DL. The effect of pudendal block on voiding after hemorrhoidectomy. Dis Colon Rectum. 2005 Mar;48(3):518-23. doi: 10.1007/s10350-004-0798-2. PMID 15875295
- [Result] Haveran LA, Sturrock PR, Sun MY, McDade J, Singla S, Paterson CA, Counihan TC. Simple harmonic scalpel hemorrhoidectomy utilizing local anesthesia combined with intravenous sedation: a safe and rapid alternative to conventional hemorrhoidectomy. Int J Colorectal Dis. 2007 Jul;22(7):801-6. doi: 10.1007/s00384-006-0242-2. Epub 2006 Nov 22. PMID 17119982